CLINICAL TRIAL: NCT03922581
Title: Primary-Care Based Mindfulness Intervention for Chronically Traumatized Individuals
Brief Title: Primary-Care Based Mindfulness Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Abigail Lott, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00104519; K23AT009713 (NIH)
Record Dates: First submitted 2019-04-18; First posted 2019-04-22 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Post Traumatic Stress Disorder; Major Depressive Disorder
Keywords: Anxiety disorders; Behavioral intervention; Psychology
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depressive Disorder, Major; Anxiety Disorders | interventions — Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Intervention Model Description: Participants will be randomized with block stratified randomization (in blocks of 20) to ensure variability in PTSD and MDD diagnosis in the two groups.
Who Masked: Outcomes Assessor
Masking Description: Staff members conducting the Clinician Administered PTSD Scale and the Mini-International Neuropsychiatric Interview will be blind to study arm assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-Based Cognitive Therapy (Experimental): Participants randomized to this study arm will receive Mindfulness-Based Cognitive Therapy (MBCT) for 8 weeks.
  Interventions: Behavioral: Mindfulness-Based Cognitive Therapy
- Wait-list Control Group (No Intervention): Participants randomized to the wait-list control study arm will be administered the study assessments while not receiving active treatment. Participants will be given the opportunity to participate in the MBCT intervention following completion of the study assessments.

INTERVENTIONS:
Behavioral: Mindfulness-Based Cognitive Therapy — The intervention consists of MBCT for the prevention of depression relapse with adaptations for discussing trauma and PTSD. Participants attend eight, weekly 90-minute group sessions involving skills training and in-class practice. Participants will return one month after the intervention has ended for a follow-up assessment.
  Arms: Mindfulness-Based Cognitive Therapy

SUMMARY:
The purpose of this study is to pilot a primary-care based mindfulness intervention for chronically traumatized African Americans screening positive for posttraumatic stress disorder (PTSD) and major depressive disorder (MDD) in primary care clinics within an urban public hospital. The study will utilize a randomized controlled trial (RCT) design along with a multi-method psychological and physiological assessment approach to establish the feasibility and acceptability of a mindfulness-based cognitive therapy (MBCT) intervention for primary care versus wait-list control in African Americans with chronic trauma exposure and comorbid PTSD and MDD. Preliminary mechanisms of action associated with MBCT including emotion dysregulation and autonomic function will be evaluated. The data collection and 8-session group intervention will take place in primary care clinics within an urban public hospital serving primarily low-income, minority individuals (>80% African American).

DETAILED DESCRIPTION:
There is significant public health burden of chronic trauma exposure in low income, predominantly ethnic minority, urban communities, which is reflected in the extraordinarily high levels of trauma-related psychiatric disorders, particularly PTSD and MDD. Despite this, limited access to behavioral health treatment and significant barriers to treatment engagement and success remain and integrating mind-body approaches in medical settings could be a critical next step in treating chronically traumatized individuals in these urban settings. This study will utilize a randomized controlled trial design along with a multi-method assessment approach to ascertain the feasibility, acceptability, and preliminary mechanisms of action and outcomes of mindfulness-based cognitive therapy versus wait-list control in 80 African Americans with chronic trauma exposure and comorbid PTSD and MDD symptoms.

Participants will be randomized to an 8-session (90 minutes each) group intervention or wait-list control. The researchers will examine the retention and follow-up rates, participants' report of acceptability and interest in the intervention, and examine barriers to treatment engagement through self-report measures and exit interviews. This study will also investigate preliminary mechanisms of action and outcomes of the mindfulness intervention in targeting emotion regulation and autonomic processes by measuring self-report of emotion dysregulation using the Difficulties in Emotion Regulation Scale and autonomic arousal to trauma cues using eSense technology to assess skin conductance during administration of Standardized Trauma Interview. Latent growth modeling will assess relative changes in emotion dysregulation and autonomic function over time through intervention and 1 month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* ability to provide informed consent
* willingness to participate in study
* self-identity as African American
* history of childhood and/or adult trauma exposure (3 total criterion A traumas)
* positive PTSD screen (PC-PTSD ≥ 3)
* positive MDD screen (PHQ-9 ≥ 5)

Exclusion Criteria:

* presence of intellectual disability, bipolar, or psychotic disorder
* presence of current substance use disorder (past 1 month)
* active suicidality

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-09-14 (Actual); Primary Completion 2023-08-18 (Actual); Study Completion 2023-08-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abigail Lott, PhD, Principal Investigator — Emory University
Locations (1):
- Grady Health System, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data collected that underlie the research results reported in the article will be available for sharing, after deidentification.
Supporting Information: Study Protocol
Time Frame: Specific data from analyses submitted for publication will be available 6 months following publication with no end date.
Access Criteria: Data will be shared with researchers who provide a methodologically sound proposal, for individual participant report meta-analysis. Specific data sharing requests should be directed to adpower@emory.edu. To gain access, requestors will need to sign a data access agreement. Data will be available indefinitely at a link to be provided.

REFERENCES:
- [Derived] Powers A, Lipschutz R, Lathan EC, Mekawi Y, Dixon HD, Bradley B, Kaslow NJ, Nugent NR. Improved Mindfulness Following Mindfulness-Based Cognitive Therapy: Results from a Pilot Randomized Controlled Trial with Trauma-Exposed Black Adults. Mindfulness (N Y). 2025;16(11):3163-3176. doi: 10.1007/s12671-025-02693-7. Epub 2025 Oct 27. PMID 41347209
- [Derived] Lathan EC, McAfee EE, Spivey BN, Garcia V, Kaslow N, Powers A. Risk for posttraumatic stress disorder symptoms by trauma type: The role of self-compassion. Psychol Trauma. 2025 Mar;17(3):603-611. doi: 10.1037/tra0001707. Epub 2024 Jul 11. PMID 38990692
- [Derived] Powers A, Lathan EC, Dixon HD, Mekawi Y, Hinrichs R, Carter S, Bradley B, Kaslow NJ. Primary care-based mindfulness intervention for posttraumatic stress disorder and depression symptoms among Black adults: A pilot feasibility and acceptability randomized controlled trial. Psychol Trauma. 2023 Jul;15(5):858-867. doi: 10.1037/tra0001390. Epub 2022 Oct 20. PMID 36265048

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from Grady Health System in Atlanta, Georgia, USA. Participant enrollment began September 14, 2018 and the final study assessment occurred on August 18, 2023.
Pre-assignment Details: Study enrollment was suspended in March 2020 due to the Coronavirus 2019 (COVID-19) pandemic. Enrollment reopened in September 2020 with a virtual intervention, rather than an in-person intervention.
Groups:
- Mindfulness-Based Cognitive Therapy: Participants randomized to receive Mindfulness-Based Cognitive Therapy (MBCT) for 8 weeks.
  Mindfulness-Based Cognitive Therapy: The intervention consists of MBCT for the prevention of depression relapse with adaptations for discussing trauma and PTSD. Participants attend eight, weekly 90-minute group sessions involving skills training and in-class practice. Participants return one month after the intervention has ended for a follow-up assessment.
- Wait-list Control Group: Participants randomized to the wait-list control study arm were administered the study assessments while not receiving active treatment. Participants were given the opportunity to participate in the MBCT intervention following completion of the study assessments.
Period: Overall Study
Arm/Group | Mindfulness-Based Cognitive Therapy | Wait-list Control Group
Started | 44 | 36
Started In-Person Intervention (Participants enrolled between September 2018 and March 2020) | 18 | 16
In-Person Intervention Participants Completing the Post-Intervention Assessment (Participants enrolled between September 2018 and March 2020) | 11 | 15
In-Person Intervention Participants Completing the Follow-up Assessment 1 Month After Intervention (Participants enrolled between September 2018 and March 2020) | 10 | 14
Started Virtual Intervention (Participants enrolled after study re-opened in September 2020) | 26 | 20
Virtual Intervention Participants Completing the Post-Intervention Assessment (Participants enrolled after study re-opened in September 2020) | 14 | 18
Virtual Intervention Participants Completing the Follow-up Assessment 1 Month After Intervention (Participants enrolled after study re-opened in September 2020) | 12 | 12
Completed | 22 | 26
Not Completed | 22 | 10
Not completed — Lost to Follow-up | 20 | 9
Not completed — Physician Decision | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- In-Person Mindfulness-Based Cognitive Therapy: Participants randomized to receive Mindfulness-Based Cognitive Therapy (MBCT) for 8 weeks. Participants enrolled between September 2018 and March 2020 received at least some of the intervention in-person.
- In-Person Wait-list Control Group: Participants randomized to the wait-list control study arm were administered the study assessments while not receiving active treatment. Participants were given the opportunity to participate in the MBCT intervention following completion of the study assessments. Participants enrolled between September 2018 and March 2020 received at least some of the intervention in-person.
- Virtual Mindfulness-Based Cognitive Therapy: Participants randomized to receive Mindfulness-Based Cognitive Therapy (MBCT) for 8 weeks. Participants enrolled after recruitment re-opened in September 2020 received the intervention virtually.
- Virtual Wait-list Control Group: Participants randomized to the wait-list control study arm were administered the study assessments while not receiving active treatment. Participants were given the opportunity to participate in the MBCT intervention following completion of the study assessments. Participants enrolled after recruitment re-opened in September 2020 received the intervention virtually.
- Total: Total of all reporting groups
Arm/Group | In-Person Mindfulness-Based Cognitive Therapy | In-Person Wait-list Control Group | Virtual Mindfulness-Based Cognitive Therapy | Virtual Wait-list Control Group | Total
Number analyzed (Participants) | 18 | 16 | 26 | 20 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.5 (12.3) | 44.3 (11.8) | 43.54 (13.78) | 45.45 (14.09) | 44.81 (12.98)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One participant in the In-Person Mindfulness-Based Cognitive Therapy study arm asked for their study data to be destroyed when they withdrew from the study.
  Participants
    number analyzed (Participants) | 17 | 16 | 26 | 20 | 79
    Female | 14 | 14 | 21 | 19 | 68
    Male | 3 | 2 | 5 | 1 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 18 | 16 | 24 | 19 | 77
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18 | 16 | 26 | 20 | 80

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Retained in Study
Description: Retention rates were assessed using session attendance. Previous mindfulness-based stress reduction (MBSR) interventions among low-income minority populations have yielded completion rates of 53-80%. Based on 80% completion rates of MBSR in primary care and 75% completion rates of MBCT both in combat vet samples and the anticipated improved accessibility through primary care, it is expected that subjects in the intervention group will evidence at least 75% retention and follow-up rates.
Time Frame: Baseline through Follow-up (1 month after the end of the 8-week intervention)
Measure: Count of Participants; unit: Participants
Groups:
- Mindfulness-Based Cognitive Therapy: Participants randomized to receive Mindfulness-Based Cognitive Therapy (MBCT) for 8 weeks.
Arm/Group | Mindfulness-Based Cognitive Therapy | Wait-list Control Group
Number analyzed (Participants) | 44 | 36
Participants | 22 | 26

2. Primary Outcome: Client Satisfaction Questionnaire (CSQ) Score
Description: Feasibility and acceptability of the Mindfulness-Based Cognitive Therapy intervention was assessed using the Client Satisfaction Questionnaire (CSQ). The CSQ is an 8-item questionnaire asking respondents to rate the quality of care they received on a scale from 1 to 4 where 1 = poor and 4 = excellent. Total raw scores range from 8 to 32 where higher values indicate greater satisfaction.
Time Frame: Week 8 (post-intervention assessment)
Population: This analysis includes participants in the MBCT study arm who completed the Post-Intervention Assessment (25 participants) and who completed this questionnaire. Three participants had missing CSQ data due to an error where the questionnaire was not administered at this time-point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Cognitive Therapy
Number analyzed (Participants) | 22
score on a scale | 30.36 (2.01)

3. Primary Outcome: Perceived Barriers to Psychological Treatment (PBPT) Scale Score
Description: Barriers to treatment was assessed using the Perceived Barriers to Psychological Treatment (PBPT) scale. The PBPT is a 25-item scale asking respondents about factors that interfere with attending weekly therapy. Items are rated on a 5-point scale where 1 = impossible to attend and 5 = not a problem. Total raw scores range from 25 to 125 where higher scores indicate low barriers regarding attending psychotherapy.
Time Frame: Week 8 (post-intervention assessment)
Population: This analysis includes participants who completed the post-intervention assessment. Two participants in the Wait-list Control Group do not have data for the PBPT due to an error in not administering the instrument.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Cognitive Therapy | Wait-list Control Group
Number analyzed (Participants) | 25 | 31
score on a scale | 48.23 (15.60) | 53.70 (18.04)

4. Primary Outcome: Difficulties in Emotion Regulation Scale (DERS) Score
Description: The Difficulties in Emotion Regulation Scale (DERS) is a 36-item instrument assessing emotion dysregulation and includes six subscales (non-acceptance of emotions, difficulty with goal-directed behavior in the presence of negative emotions, difficulty controlling impulses in the presence of negative emotions, lack of awareness of emotions, limited use of effective emotion regulation strategies, and lack of understanding of emotions). Responses are scaled from 1 (almost never) to 5 (almost always). Total raw scores range from 36 to 180; certain items are reverse scored so that higher scores indicate increased difficulty with emotion regulation.
Time Frame: Baseline, Weeks 3, 5, 7, 8 (post-intervention assessment), and Follow-up (1 month after the end of the intervention)
Population: One participant in MBCT requested all data removed so baseline score was unavailable; 1 participant in MBCT and 2 participants in Wait-list Control (WLC) had multiple missing self-report measures at baseline due to interviewer error. Missing data at Weeks 3, 5, and 7 were related to a participant not present at group or unable to be reached for the assessment component. The DERS was not administered to the WLC group at Weeks 3 and 7.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Cognitive Therapy | Wait-list Control Group
Number analyzed (Participants) | 42 | 34
score on a scale
  Baseline | 78.05 (21.09) | 83.77 (23.60)
  Week 3: number analyzed (Participants) | 24 | 0
  Week 3 | 77.08 (20.78) |
  Week 5: number analyzed (Participants) | 26 | 28
  Week 5 | 73.46 (25.17) | 83.03 (25.71)
  Week 7: number analyzed (Participants) | 17 | 0
  Week 7 | 73.17 (21.70) |
  Week 8: number analyzed (Participants) | 25 | 29
  Week 8 | 71.24 (26.55) | 73.55 (24.36)
  Follow-up one month after end of intervention: number analyzed (Participants) | 21 | 26
  Follow-up one month after end of intervention | 73.00 (25.70) | 80.56 (29.78)

5. Primary Outcome: Number of Participants Reporting Change in Experience of Emotions or Handling Stressful Situations in Post-group Follow-up Questionnaire
Description: Participants randomized to the MBCT intervention completed an open-ended, follow-up questionnaire designed to assess feelings and changes experienced from participation in the intervention. Participants were asked "Have you noticed any changes in how you experience emotions or handle stressful situations?". Responses were given in text form rather than on a pre-set scale, and were then categorized as positive change, no change, or negative change.
Time Frame: Week 8 (post-intervention assessment)
Population: This analysis includes participants receiving the MBCT intervention, either in-person or virtually, who attended the post-intervention assessment and responded to this question.
Measure: Count of Participants; unit: Participants
Arm/Group | In-Person Mindfulness-Based Cognitive Therapy | Virtual Mindfulness-Based Cognitive Therapy
Number analyzed (Participants) | 15 | 13
Participants
  Positive change | 15 | 11
  No change | 0 | 2
  Negative change | 0 | 0

6. Primary Outcome: Skin Conductance Among In-Person Intervention Participants
Description: Skin conductance (SC) response was measured among participants receiving the in-person intervention using a mobile SC device, eSense (Mindfield Biosystems). Continuous recording of SC is measured with electrodes on hands and data is transmitted through the eSense app. Using the PhenX Toolkit protocol, a two minute baseline measure of SC will be obtained and then SC levels were measured during administration of the Standardized Trauma Interview immediately following to determine physiological reactivity to trauma stimuli. SC response is calculated by subtracting SC level at the end of baseline recording (average of last 30 seconds) from the maximum SC level value during the trauma interview.
Time Frame: Baseline, Week 8 (post-intervention assessment)
Population: 8 MBCT and 8 WLC participants do not have usable baseline data due to a missing measurement, noise/error in output, iPad malfunction, or request for data removal. 2 MBCT participants and 7 WLC participants do not have Week 8 data because it was unusable due to noise/error in output. 3 MBCT participants and 1 WLC participants missed SC data collection at Week 8 due to onset of the COVID-19 pandemic and 2 WLC participants were missing SC data collection at Week 8 due to iPad malfunction.
Measure: Mean (Standard Deviation); unit: µSiemens (µS)
Arm/Group | Mindfulness-Based Cognitive Therapy | Wait-list Control Group
Number analyzed (Participants) | 10 | 8
µSiemens (µS)
  Baseline | 1.39 (1.60) | 1.29 (1.77)
  Week 8: number analyzed (Participants) | 6 | 5
  Week 8 | 1.07 (1.22) | 0.62 (0.64)

7. Secondary Outcome: Number of Participants With PTSD by Primary Care PTSD Screen (PC-PTSD) Determination
Description: The Primary Care PTSD Screen (PC-PTSD) is a 5-item screen designed for use in primary care used to assess for presence of PTSD symptoms and serve as PTSD screener. Respondents answer "yes" or "no" to each question and an individual is considered to have PTSD if they respond with "yes" to at least 3 of the 5 questions.
Time Frame: Baseline, Week 8 (post-intervention assessment), Follow-up (1 month after the end of the intervention)
Population: 1 participant in the MBCT condition requested all data removed so baseline score was unavailable. Additional missing data at Week 8 and Follow-up were due to interviewer error in not asking all the self-report questions or if a participant ran out of time and ended the assessment early and was unable to be reached at a later time to finish the assessment battery.
Measure: Count of Participants; unit: Participants
Arm/Group | Mindfulness-Based Cognitive Therapy | Wait-list Control Group
Number analyzed (Participants) | 43 | 36
Participants
  Baseline | 43 | 36
  Week 8: number analyzed (Participants) | 23 | 28
  Week 8 | 16 | 21
  Follow-up: number analyzed (Participants) | 20 | 23
  Follow-up | 10 | 15

8. Secondary Outcome: Patient Health Questionnaire-9 (PHQ-9) Score
Description: The Patient Health Questionnaire-9 (PHQ-9) will assess for presence of depressive symptoms and serve as a major depressive disorder (MDD) screening tool. The PHQ-9 is a 9-item tool that asks respondents to indicate how frequently they have felt symptoms of depression on a scale of 0 to 3 where 0 = not at all and 3 = nearly every day. Total scores range from 0 to 27, where higher scores indicate worse depression.
Time Frame: Baseline, Week 8 (post-intervention assessment), Follow-up (1 month after the end of the intervention)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Cognitive Therapy | Wait-list Control Group
Number analyzed (Participants) | 43 | 36
score on a scale
  Baseline | 17.35 (4.71) | 18.67 (4.06)
  Week 8: number analyzed (Participants) | 23 | 28
  Week 8 | 13.30 (8.09) | 13.64 (6.17)
  Follow-up: number analyzed (Participants) | 20 | 23
  Follow-up | 12.47 (6.95) | 14.22 (6.03)

9. Secondary Outcome: PTSD Checklist for Diagnostic and Statistical Manual of Mental Disorders (DSM)-5 (PCL-5) Score
Description: The PCL-5 is a 20-item questionnaire asking respondents to report how much they have been bothered by problems in the past month on a scale of 0 (not at all) to 4 (extremely). Total scores range from 0 to 80 where higher scores indicate increased difficulty with responses to stressful experiences.
Time Frame: Baseline, Week 8 (post-intervention assessment)
Population: 1 participant in the MBCT condition requested all data removed so baseline score was unavailable. Baseline data for 1 MBCT participant and 1 WLC participant was missing due to interviewer error. Additional missing data at Week 8 and Follow-up were due to interviewer error in not asking all the self-report questions or if a participant ran out of time and ended the assessment early and was unable to be reached at a later time to finish the assessment battery.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Cognitive Therapy | Wait-list Control Group
Number analyzed (Participants) | 42 | 35
score on a scale
  Baseline | 49.12 (14.07) | 54.86 (11.73)
  Week 8: number analyzed (Participants) | 24 | 27
  Week 8 | 34.91 (20.17) | 37.41 (18.60)

10. Secondary Outcome: Beck Depression Inventory-II (BDI-II) Score
Description: The BDI-II is a 21-item instrument asking respondents to indicate how much they are bothered by negative feelings. Responses are on a scale of 0 to 3 where 0 = the problematic feeling is not present and 3 = the feeling is very strong. Total scores range from 0 to 63, where high scores indicate worse problems with negative feelings.
Time Frame: Baseline, Week 8 (post-intervention assessment)
Population: 1 participant in the MBCT condition requested all data removed so baseline score was unavailable. Baseline data for 3 MBCT participants were also missing due to interviewer error. Additional missing data at Week 8 were due to interviewer error in not asking all the self-report questions or if a participant ran out of time and ended the assessment early and was unable to be reached at a later time to finish the assessment battery.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Cognitive Therapy | Wait-list Control Group
Number analyzed (Participants) | 40 | 36
score on a scale
  Baseline | 33.80 (11.13) | 36.39 (10.42)
  Week 8: number analyzed (Participants) | 24 | 26
  Week 8 | 24.94 (14.25) | 25.16 (13.81)

11. Secondary Outcome: Number of Participants Diagnosed With PTSD Using the Clinician Administered PTSD Scale
Description: The Clinician Administered PTSD Scale is a semi-structured interview used for diagnosing PTSD. The number of participants diagnosed with PTSD pre- and post-intervention will be compared between study arms.
Time Frame: Baseline, Week 8 (post-intervention assessment)
Population: 1 participant in the MBCT condition requested all data removed so baseline score was unavailable.
Measure: Count of Participants; unit: Participants
Arm/Group | Mindfulness-Based Cognitive Therapy | Wait-list Control Group
Number analyzed (Participants) | 43 | 36
Participants
  Baseline | 32 | 21
  Week 8: number analyzed (Participants) | 25 | 33
  Week 8 | 9 | 21

12. Secondary Outcome: Mini International Neuropsychiatric Interview (MINI) MDD Determination
Description: The Mini International Neuropsychiatric Interview (MINI) is a semi-structured interview used for diagnosing MDD. The number of participants diagnosed with MDD pre- and post-intervention will be compared between study arms.
Time Frame: Baseline, Week 8 (post-intervention assessment)
Population: 1 participant in the MBCT condition requested all data removed so baseline score was unavailable.
Measure: Count of Participants; unit: Participants
Arm/Group | Mindfulness-Based Cognitive Therapy | Wait-list Control Group
Number analyzed (Participants) | 43 | 36
Participants
  Baseline | 26 | 23
  Week 8: number analyzed (Participants) | 25 | 33
  Week 8 | 12 | 16

13. Secondary Outcome: Five Facet Mindfulness Questionnaire Score
Description: The Five Facet Mindfulness Questionnaire is a 39-item instrument assessing mindfulness, and includes five facets (observing, describing, acting with awareness, non-judging of inner experience, and non-reactivity to inner experience). Participants respond to each item on a scale of 1 to 5 where 1 = the statement is never or very rarely true for them and 5 = the statement is very often or always true. Total raw scores range from 39 to 195; certain items are reverse scored so that higher scores indicate increased mindfulness.
Time Frame: Baseline, Week 8 (post-intervention assessment), Follow-up (1 month after the end of the intervention)
Population: 1 participant in the MBCT condition requested all data removed so baseline score was unavailable. Additional missing data at Baseline, and Week 8 were due to interviewer error in not asking all the self-report questions or if a participant ran out of time and ended the assessment early and was unable to be reached at a later time to finish the assessment battery.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Cognitive Therapy | Wait-list Control Group
Number analyzed (Participants) | 42 | 31
score on a scale
  Baseline | 119.81 (19.82) | 122.39 (21.40)
  Week 8: number analyzed (Participants) | 26 | 29
  Week 8 | 124.35 (30.68) | 122.46 (22.16)
  Follow-up: number analyzed (Participants) | 22 | 26
  Follow-up | 130.14 (24.13) | 121.15 (24.21)

14. Secondary Outcome: Self Compassion Scale, Short Form Score
Description: The Self Compassion Scale is a 12-item instrument assessing how respondents typically act towards themselves during difficult times. Items are answered on a scale of 1 to 5 where 1 = almost never and 5 = almost always. Total scores range from 12 to 60; certain items are reversed scored so that higher scores indicate increased self compassion.
Time Frame: Baseline, Week 8 (post-intervention assessment), Follow-up (1 month after the end of the intervention)
Population: 1 participant in the MBCT condition requested all data removed so baseline score was unavailable. Additional missing data at Baseline, Week 8 and Follow-up were due to interviewer error in not asking all the self-report questions or if a participant ran out of time and ended the assessment early and was unable to be reached at a later time to finish the assessment battery.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Cognitive Therapy | Wait-list Control Group
Number analyzed (Participants) | 39 | 29
score on a scale
  Baseline | 31.44 (8.01) | 32.45 (8.15)
  Week 8: number analyzed (Participants) | 24 | 28
  Week 8 | 35.42 (10.86) | 33.68 (12.59)
  Follow-up: number analyzed (Participants) | 20 | 25
  Follow-up | 34.65 (10.86) | 34.04 (12.59)

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected at all assessment and session visits with study participants following baseline assessment and continued through the follow-up assessment occurring one month after the end of the intervention (or WLC condition). All adverse event data during study participation is included below. WLC participants were eligible to participate in the MBCT group after study participation but adverse events were not monitored for those individuals post study completion.
Arm/Group | Mindfulness-Based Cognitive Therapy | Wait-list Control Group
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/36
Other Adverse Events (participants affected / at risk) | 11/44 | 3/36
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mindfulness-Based Cognitive Therapy (N=44) | Wait-list Control Group (N=36)
Mood symptom increase (Psychiatric disorders) | 2 | 2
Anxiety symptom increase (Psychiatric disorders) | 1 | 0
Coronavirus Disease 2019 (COVID-19) (Infections and infestations) | 1 | 0
Work related physical injury (Injury, poisoning and procedural complications) | 1 | 0
Prolonged menstrual bleeding related to birth control pill (Reproductive system and breast disorders) | 1 | 0
Stitches on toe (Surgical and medical procedures) | 1 | 0
Lump in armpit (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Worsening arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Worsening chronic pain (General disorders) | 2 | 0
Headache (General disorders) | 1 | 0
Hernia (Musculoskeletal and connective tissue disorders) | 1 | 0
Eye dryness/irritation (Eye disorders) | 1 | 0
Chest pain (Cardiac disorders) | 1 | 0
Chronic liver dysfunction diagnosis (Hepatobiliary disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-01-21): https://cdn.clinicaltrials.gov/large-docs/81/NCT03922581/Prot_SAP_001.pdf
  • Informed Consent Form (2022-01-27): https://cdn.clinicaltrials.gov/large-docs/81/NCT03922581/ICF_000.pdf